CLINICAL TRIAL: NCT01035853
Title: Sino-nasal Inhalation of Colistin Via the Pari Sinus Nebulizer in Patients With Cystic Fibrosis and Colonization of the Upper Airways With Pseudomonas Aeruginosa
Brief Title: Sino-nasal Inhalation of Colistin in Patients With Cystic Fibrosis and Pseudomonas Aeruginosa Colonization
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Jena (Other)
Responsible Party: Principal Investigator, PD Dr. Jochen G. Mainz, PD Dr., University of Jena
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: colistin nasal cf pilot
Record Dates: First submitted 2009-12-17; First posted 2009-12-21 (Estimated); Last update posted 2013-03-21 (Estimated); Status verified 2013-03

CONDITIONS: Cystic Fibrosis; Pseudomonas Aeruginosa
MeSH Terms: conditions — Cystic Fibrosis; Pseudomonas Infections | interventions — Colistin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Colistin — Sino-Nasal inhalation, approximately 1 ml / day in each nostril

SUMMARY:
The purpose of this study is to determine whether the nasal inhalation of Colistin is effective to decrease the Pseudomonas aeruginosa bacterial count in the nasal lavage fluid.

ELIGIBILITY:
Inclusion Criteria:

* subject has a confirmed diagnosis of cystic fibrosis
* detection of P. aeruginosa in nasal lavage (culture) with chronic P.a. colonization of the lung (from day -28)
* informed consent of the patients or parents
* subject >= 6 years
* subject is able to comply with the inhalation procedures and nasal lavage procedures scheduled in the protocol
* women of childbearing potential are only included into the study, if they are using an effective method of birth control during the protocol

Exclusion Criteria:

* subject has a critical condition defined as: forced expiratory volume at one second < 30% and / or arterial oxygen saturation < 93% without O2-substitution; need of O2-substitution
* subject had an ear, nose, and throat surgery within 3 months prior to study
* subject shows signs of nasal bleeding
* subject has an ear drum perforation
* subject had an acute rhinosinusitis or a pulmonary exacerbation at study entry with need of additional systemic antibiotic therapy against pseudomonas aeruginosa
* subject is unlikely to comply with the procedures scheduled in the protocol
* subject has a known allergic reaction to the medication
* subject is pregnant or breastfeeding
* subject participates in another clinical trial within 30 days prior to study entry or 30 days after end of the study.
* systemic (oral or intravenous) antibiotic treatment against P.a. 14 days prior to the inclusion and during the study

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Decrease of Pseudomonas aeruginosa in Nasal lavage fluid | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Mainz, M.D., Study Chair — University of Jena, Children's hospital
Locations (3):
- Germany (3):
  - Universitäts-Kinderklinik, Tübingen, Baden-Würtemberg
  - Mukoviszidosezentrum der Friedrich-Schiller-Universität, Jena, Thuringia
  - CF-Zentrum, Hamburg